CLINICAL TRIAL: NCT00054457
Title: A Phase II Study Of Docetaxel And Capecitabine In Patients With Measurable Metastatic Adenocarcinoma Of The Stomach And Gastroesophageal Junction
Brief Title: Docetaxel and Capecitabine in Treating Patients With Metastatic Cancer of the Stomach or Gastroesophageal Junction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N0242; NCI-2012-02517 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000270681 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-12

CONDITIONS: Esophageal Cancer; Gastric Cancer
Keywords: adenocarcinoma of the stomach; adenocarcinoma of the esophagus; stage IV gastric cancer; recurrent gastric cancer; stage IV esophageal cancer; recurrent esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Adenocarcinoma Of Esophagus | interventions — Capecitabine; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- docetaxel + capecitabine (Experimental): Patients receive docetaxel IV over 1 hour on day 1 and oral capecitabine twice daily on days 1-14. Courses repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Quality of life is assessed at baseline, at each tumor measurement, and at the end of treatment.
  Patients are followed every 3 months until disease progression and then every 6 months until 3 years from registration.
  Interventions: Drug: capecitabine; Drug: docetaxel

INTERVENTIONS:
Drug: capecitabine
Drug: docetaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study of the effectiveness of combining docetaxel with capecitabine in treating patients who have metastatic cancer of the stomach or gastroesophageal junction.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the objective tumor response rate in patients with metastatic gastric or gastroesophageal junction adenocarcinoma treated with docetaxel and capecitabine.
* Determine the time to progression in patients treated with this regimen.
* Determine the overall survival in patients treated with this regimen.
* Determine the toxic effects of this regimen in these patients.
* Determine whether interleukin-1 polymorphisms are present among patients who have weight loss vs no weight loss, and their relationship to a poor prognosis.
* Assess the quality of life and swallowing uniscale during chemotherapy in these patients.

OUTLINE: Patients receive docetaxel IV over 1 hour on day 1 and oral capecitabine twice daily on days 1-14. Courses repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, at each tumor measurement, and at the end of treatment.

Patients are followed every 3 months until disease progression and then every 6 months until 3 years from registration.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the stomach or gastroesophageal junction
* Deemed unresectable and not a candidate for potentially curative treatment (e.g., surgical resection or combined modality therapy)

  * At least 4 weeks since prior abdominal exploration with resection (3 weeks without resection)
  * No other more conventional forms of therapy available with a reasonable chance of cure or significant palliation
* Measurable disease*

  * The following are not considered measurable disease:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusion
    * Lymphangitis cutis/pulmonis
    * Abdominal masses that are not confirmed and followed by imaging
    * Cystic lesions NOTE: *Patients having only lesions measuring ≥ 1 cm to < 2 cm must use spiral CT scan for all tumor assessments.
* No untreated or treated but symptomatic CNS metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 12 weeks

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than upper limit of normal (ULN)
* AST no greater than 2.5 times ULN if alkaline phosphatase is less than ULN OR
* Alkaline phosphatase no greater than 4 times ULN if AST less than ULN

Renal

* Creatinine normal
* Creatinine clearance at least 60 mL/min

Cardiovascular

* No New York Heart Association class III or IV heart disease

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Ability to swallow capecitabine
* No prior anaphylactic reaction to any taxane
* No prior severe reaction to fluoropyrimidine
* No prior poor tolerance to capecitabine
* No known sensitivity or poor tolerance to fluorouracil
* No known dihydropyrimidine dehydrogenase deficiency
* No uncontrolled infection
* No uncontrolled seizure disorder
* No chronic debilitating disease
* No peripheral neuropathy of any etiology greater than grade 1
* No diabetes mellitus
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell carcinoma or adequately treated noninvasive carcinoma

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior immunotherapy or biologic therapy for recurrent or metastatic disease
* No concurrent biologic therapy

Chemotherapy

* No prior chemotherapy for recurrent or metastatic disease except for the following:

  * Adjuvant chemotherapy after complete resection of the original tumor
  * Neoadjuvant chemotherapy followed by surgical resection of the original tumor
* No other concurrent chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy except for the following:

  * Adjuvant radiotherapy after complete resection of the original tumor
  * Neoadjuvant radiotherapy followed by surgical resection of the original tumor
* No prior radiotherapy to 25% or more of the bone marrow
* More than 4 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery

* See Disease Characteristics
* No prior organ allograft

Other

* No concurrent brivudine or sorivudine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2003-09; Primary Completion 2007-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Proportion of successes | Up to 3.5 years

SECONDARY OUTCOMES:
Survival time | Up to 3.5 years
Time to disease progression | Up to 3.5 years
Duration of response | Up to 3.5 years
Time to treatment failure | Up to 3.5 years
Quality of life as measured by the LASA, FACT-E and Patient Uniscale Swallowing questionnaires | Up to 3.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Aminah Jatoi, MD, Study Chair — Mayo Clinic
Locations (28):
- United States (28):
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota

REFERENCES:
- [Background] Jatoi A, Foster NR, Egner JR, Burch PA, Stella PJ, Rubin J, Dakhil SR, Sargent DJ, Murphy BR, Alberts SR. Older versus younger patients with metastatic adenocarcinoma of the esophagus, gastroesophageal junction, and stomach: a pooled analysis of eight consecutive North Central Cancer Treatment Group (NCCTG) trials. Int J Oncol. 2010 Mar;36(3):601-6. doi: 10.3892/ijo_00000535. PMID 20126980
- [Result] Jatoi A, Nguyen PL, Foster N, Sun D, Stella PJ, Campbell M, Tschetter LK, Dakhil SR, Mailliard JA, Nikcevich DA. Interleukin-1 genetic polymorphisms and their relationship to the cancer anorexia/weight loss syndrome in metastatic gastric and gastroesophageal junction adenocarcinoma. J Support Oncol. 2007 Jan;5(1):41-6. PMID 17265786
- [Result] Giordano KF, Jatoi A, Stella PJ, Foster N, Tschetter LK, Alberts SR, Dakhil SR, Mailliard JA, Flynn PJ, Nikcevich DA; North Central Cancer Treatment Group. Docetaxel and capecitabine in patients with metastatic adenocarcinoma of the stomach and gastroesophageal junction: a phase II study from the North Central Cancer Treatment Group. Ann Oncol. 2006 Apr;17(4):652-6. doi: 10.1093/annonc/mdl005. Epub 2006 Feb 23. PMID 16497828